CLINICAL TRIAL: NCT06050057
Title: Possibilities of Surgical Treatment of Adrenal Diseases: Comparison of Laparoscopic and Robotic-assisted Adrenalectomy-a Prospective Study
Brief Title: Surgical Treatment of Adrenal Diseases- Laparoscopic vs. Robotic-assisted Adrenalectomy
Status: Recruiting | Type: Observational
Sponsor: University Hospital Olomouc (Other)
Collaborators: University Hospital Ostrava (Other); Tomas Bata Hospital, Czech Republic (Other); General University Hospital, Prague (Other); University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Natalia Wiesner, Head of the urological clinic, MUDr. Igor Hartmann Ph.D., University Hospital Olomouc
Other Study IDs: FNOL 122/23
Record Dates: First submitted 2023-09-04; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Adrenal Tumor; Adrenal Disease; Adrenal Mass; Adrenalectomy; Status; Adrenal Hyperplasia; Adrenal Gland Metastasis; Adrenal Cortex Diseases; Pheochromocytoma; Cushing Syndrome; Conn Adenoma; Adrenocortical Carcinoma; Adrenocortical Adenoma; Adrenocortical Tumor
Keywords: Adrenal Tumor; Pheochromocytoma; Conn Adenoma; Cushing Syndrome; Adrenalectomy; Laparoscopic surgery; da Vinci surgical system
MeSH Terms: conditions — Adrenal Gland Neoplasms; Adrenal Gland Diseases; Adrenal Hyperplasia, Congenital; Adrenal Cortex Diseases; Pheochromocytoma; Cushing Syndrome; Adrenocortical Adenoma; Adrenocortical Carcinoma; Adrenal Cortex Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this multicenter, observational, analytic, randomized clinical trial is to analyze the laparoscopic and robot-assisted method in the surgical treatment of patients with adrenal diseases. The main question it aims to answer are:

1. to find the superiority of one the the surgical method mentioned above
2. to compare the quality of life in patients with adrenal mass before surgery and after laparoscopic or robotic-assisted adrenalectomy.

ELIGIBILITY:
Inclusion Criteria:

* Indicated adrenalectomy based on endocrinological and imaging examination.
* Written consent to participate in the study.

Exclusion Criteria:

* Simultaneous bilateral adrenalectomy.
* Adrenal expansion > 12 cm.
* Suspected malignant adrenal tumor with infiltrative growth or tumor venous thrombus according to imaging examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for adrenalectomy based on endocrinological and imaging examination. All patients older than 18 years who met the clinical criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-03 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Initial examination 1 | 1 day
  Initial examination by a urologist and indication for the surgery.
Initial examination 2 | 1 day
  Sampling of biological material: Hemoglobin g/l
Surgical period 1 | 1 day
  Measuring the operation time in minutes.
Surgical period 2 | 1 day
  Measuring the blood loss in milliliters (ml).
Surgical period 3 | 1 day
  Record the need for conversion to open surgery.
Surgical period 4 | 1 day
  Record the surgical complications.
Surgical period 5 | 1 day
  The consumption of special surgical instruments.
Perioperative period 1 | from 3- 7 days
  Perioperatively, the length of stay in the ICU in days.
Perioperative period 2 | from 3- 7 days
  Perioperatively, total hospitalization time in days
Perioperative period 3 | from 3- 7 days
  Perioperatively, blood loss from the drain in mililiters (ml).
Perioperative period 4 | from 3- 7 days
  Perioperatively, time to remove the abdominal drain in days.
Perioperative period 5 | from 3- 7 days
  Perioperatively, need for blood substitutes.
Perioperative period 6 | from 3- 7 days
  Perioperatively, number of forced surgical revisions.
Perioperative period 7 | from 3- 7 days
  Perioperatively, consumption of analgesics during the hospitalization.
First post-operative check-up 1 | 1 day of examination, 14- 20 days from the surgery
  First postoperative visit (14th to 20th postoperative day), sampling of biological material: Hemoglobin g/l
First post-operative check-up 2 | 1 day of examination, 14- 20 days from the surgery
  First postoperative visit (14th to 20th postoperative day)- an analysis of perioperative and early postoperative complications according to the Dindo Clavien classification
First post-operative check-up 3 | 1 day of examination, 14- 20 days from the surgery
  First postoperative visit (14th to 20th postoperative day)- necessary hospitalizations and operative revisions.
Second post-operative check-up 1 | 1 day of examination, 85-100 days from the surgery
  Second postoperative visit (85th to 100th postoperative day)- an analysis of late postoperative complications according to the Dindo Clavien classification.
Second post-operative check-up 2 | 1 day of examination, 85-100 days from the surgery
  Second postoperative visit (85th to 100th postoperative day)- necessary hospitalizations and operative revisions

CONTACTS AND LOCATIONS:
Overall Officials: MUDr. Igor Hartmann Ph.D., Study Chair — Dpt. of Urology, University hospital Olomouc
Locations (1):
- University hospital Olomouc, Olomouc, Czechia